CLINICAL TRIAL: NCT03173430
Title: Pilot Study of Blinatumomab in Combination With Salvage Autologous Stem Cell Transplantation for Patients With Refractory Multiple Myeloma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI decided to close study due to slow accrual.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 56416
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): An evaluable subject is any subject who completes two 28-day cycles of blinatumomab or discontinues blinatumomab after completion of less than one cycle due to toxicity.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab (Blincyto), an anti-CD19/anti-CD3 bi-specific T cell engager

SUMMARY:
This study involves receiving blinatumomab after high-dose melphalan and ASCT for multiple myeloma. The main purpose of this study is to: - To determine whether blinatumomab is safe and feasible to administer after ASCT in patients with advanced multiple myeloma. - To assess how long multiple myeloma remains under control when blinatumomab is administered after second ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have undergone a prior ASCT for multiple myeloma and have progressed within 365 days of stem cell infusion. Progression is defined according to IMWG criteria49.

  * Prior ASCT must have utilized melphalan conditioning at a dose of 200 mg/m2.
  * Patients who underwent syngeneic transplant (i.e., transplant from an identical twin donor) rather than autologous transplant are eligible if syngeneic stem cells are available for use in the salvage transplant and syngeneic transplant will be considered equivalent to ASCT for the purposes of these inclusion/exclusion criteria.
  * Patients in whom first progression is identified between days 366 and 450 (inclusive) after ASCT will be eligible if progression is identified on their first evaluation for progression in this window and if they had not been evaluated between days 270 and 365 for progression. This clause is to account for practice patterns in which patients otherwise doing well are monitored infrequently (every 3-6 months) for relapse after they recover from their first ASCT. This will allow infrequently monitored patients to be included if progression is identified on their "12 month follow-up evaluation" if this appointment happens to be scheduled just outside the 365-day post-ASCT window.
  * There is no requirement that patients must enroll within 365 days of prior ASCT, and patients may be treated with other agents, including experimental agents, following relapse/progression after prior ASCT before enrollment on this study.

    * Subjects must have received as part of their initial therapy for multiple myeloma, prior to first ASCT, a regimen containing either bortezomib or lenalidomide.
* Subjects must have signed written, informed consent.
* Subjects must be ≥ 18 and ≤ 70 years of age.
* Subjects must have adequate vital organ function to undertake ASCT, defined as the following:

  * Estimated or measured creatinine clearance of ≥60 mL/min. CKD-EPI equation will be used for estimation of creatinine clearance (http://www.kidney.org/professionals/kdoqi/gfr_calculator).
  * SGOT ≤ 3x the upper limit of normal and total bilirubin ≤ 2.0 mg/dl (except for patients in whom hyperbilirubinemia is attributed to Gilbert's syndrome).
  * Left ventricular ejection fraction ≥45% as measured by echocardiography or MUGA scan.
  * Adequate pulmonary function with FEV1, FVC, TLC, and DLCO (after appropriate adjustment for lung volume and hemoglobin concentration) ≥40% of predicted values.
  * Non-hematologic toxicities from prior therapies must have recovered to grade ≤2 according to CTCAE 4.0 criteria or the subject's prior baseline.
* Subjects must have measurable disease, as defined in the IMWG response criteria49, on study entry.
* Subjects must have an ECOG performance status of 0-2 unless a higher performance status is due solely to bone pain.
* Subjects must have stored in usable condition for second ASCT, as judged by the principal investigator, ≥3x106 CD34+ cells per kg of body weight (either autologous or syngeneic) stored in at least two bags such that after administration of the minimum dose of 2 x 106 CD34+ cells/kg required on this protocol that a separate aliquot of at least 1 x 106 CD34+ cells/kg remains for rescue infusion in the event of graft failure.
* Subjects must agree not to attempt to become pregnant or impregnate others (e.g., through sexual intercourse or sperm donation) between enrollment and completion of blinatumomab therapy. Sexually active subjects with reproductive potential must agree during the study to utilize a reliable method of contraception, which may include condoms (male or female), diaphragm or cervical cap with spermicide, intrauterine device, or hormonal contraceptive. Acceptable documentation of the absence of reproductive potential may consist of any one of the following: (1) physician report/letter, (2) operative report or other source documentation of surgical sterilization, (3) laboratory report of azospermia (required to document successful vasectomy), (4) follicle stimulating hormone measurement elevated in the menopausal range.
* Due to the potential for neurological events, including seizures, while receiving blinatumomab, subjects must be willing and able to refrain from driving and engaging in hazardous occupations or activities such as operating heavy or potentially dangerous machinery during the periods of blinatumomab infusion.

Exclusion Criteria:

* Pregnant or lactating. Female subjects of reproductive potential (women who have reached menarche and who have had menses within the preceding 24 months or have not undergone hysterectomy or bilateral oophorectomy) must have a negative serum pregnancy test performed at the time of screening.
* Active and uncontrolled infection
* Positive serum testing for hepatitis B core antibody or hepatitis B surface antigen.
* Evidence of active hepatitis C or HIV infection (positive serology with appropriate positive confirmatory testing, such as nucleic acid-based testing).
* Any condition that would preclude participation as outlined in the judgment of the principal investigator.
* Prior allogeneic stem cell transplantation.
* Prior receipt of >1 autologous stem cell transplantation.
* Clinically significant CNS pathology, including documented or suspected CNS myeloma. Clinically insignificant clinical examination findings or imaging abnormalities (e.g., age-related changes) should not be cause for exclusions of potential subjects.
* Class III/IV cardiovascular disability according to the New York Heart Association Classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Garfall, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States